CLINICAL TRIAL: NCT04635267
Title: Effects of Extravascular Lung Water on Prone Position Efficacy in Patients With Acute Respiratory Distress Syndrome
Brief Title: Effects of Extravascular Lung Water on Prone Position Efficacy in Patients With ARDS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bicetre Hospital (Other)
Responsible Party: Principal Investigator, Christopher Lai, doctor, Bicetre Hospital
Other Study IDs: 2020-A03094-35
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Respiratory Distress Syndrome in Adult or Child
Keywords: ARDS; Prone Position; Extravascular lung water; Lung recruitment
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with ARDS
  Interventions: Other: Prone position in patients with ARDS

INTERVENTIONS:
Other: Prone position in patients with ARDS — Transpulmonary thermodilution, arterial blood gas and recruitment/inflation calculation will be made every 8 hours: at baseline (just before prone position), after eight hours of prone position, after 16 hours of prone position (end of prone position), after 24 hours ( 8 hours after the end of prone position).

SUMMARY:
The study will investigate the influence that extravascular lung water index (EVLWi) could have on the efficacy and persistance of efficacy of prone position in patients with acute respiratory distress syndrome.

Prone position will increase blood oxygenation in 75% of the cases and will be persistant in half of the cases. Unfortunately, no clinical criteria has been found correlated with efficacy. The quantity of lung edema, with increased lung weight, could be a determinant factor of efficacy and the persistance of the efficacy. EVLWi, assessed with the PiCCO2 device, reflects the quantity of fluid accumulated in interstitial and alveolar spaces.

The hypothesis is that patients with higher EVLWi will have less efficacy of prone position in oxygenation and also that the beneficial effects of prone position will last shorter compared to patients with lower EVLWi.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Presence of acute respiratory distress syndrome
* Decision to perform prone position according to the physician in charge of the patient
* Hemodynamic monitoring with a PiCCO2 device (Pulsion Medical Systems, Feldkirchen, Allemagne)

Exclusion Criteria:

* Absence of affiliation to the French Sociale security
* Patient under a tutelage measure or placed under judicial protection
* Known pregnancy
* Currently receiving ECMO therapy

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with moderate-to-severe ARDS in whom prone positioning is deemed necessary
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between extravascular lung water index (EVLWi) just before prone position (baseline) and the time course of the partial arterial pressure in oxygen over inspired fraction of oxygen (PaO2/FiO2) ratio during prone position. | up to 24 hours
  EVLWi is the amount of water contained in the lungs outside the pulmonary vasculature. It can be measured using the transpulmonary thermodilution technique with the PiCCO2 device (Pulsion Medical Systems, Feldkirchen, Germany)

SECONDARY OUTCOMES:
Correlation between extravascular lung water index (EVLWi) just before prone position (baseline) and the time course of the recruitment/inflation ratio during prone position. | up to 24 hours
  recruitment/inflation ratio is a validated method to characterize the lung recruitability with high positive expiratory pressure, at the bedside of patients with ARDS
Correlation between extravascular lung water index (EVLWi) at the end of prone position and the time course of the partial arterial pressure in oxygen over inspired fraction of oxygen (PaO2/FiO2) ratio in the next eight hours after prone position | up to 24 hours
  EVLWi is the amount of water contained in the lungs outside the pulmonary vasculature. It can be measured using the transpulmonary thermodilution technique with the PiCCO2 device (Pulsion Medical Systems, Feldkirchen, Germany)
Correlation between extravascular lung water index (EVLWi) at the end of prone position and the time course of the recruitment/inflation ratio in the next eight hours after prone position. | up to 24 hours
  recruitment/inflation ratio is a validated method to characterize the lung recruitability with high positive expiratory pressure, at the bedside of patients with ARDS

IPD SHARING:
Plan to Share IPD: Undecided